CLINICAL TRIAL: NCT06236646
Title: Effects of Thai Dance With Twenty-five Squares on Cerebrovascular and Cognitive Function in Elderly With Mild Cognitive Impairment
Brief Title: Effects of Thai Dance With Twenty-five Squares in Elderly With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wannaporn Tongtako, Ph.D., Principal investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EX PHYSIO SPSC 9
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Mild Cognitive Impairment
Keywords: aerobic exercise; elderly; mild cognitive impairment; cerebrovascular; respiratory function
MeSH Terms: conditions — Cognitive Dysfunction; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thai dance with twenty-five squares (TDT) (Experimental): The participants received a Thai dance with twenty-five squares (TDT) program 3 days/week, 12 weeks. This training comprises 10 minutes of warm up, following by 40 minutes of exercise at 40-50% of heart rate reserve at week 1-4, 50-60% of heart rate reserve at week 5-8, and 60-70% of heart rate reserve at week 9-12, 5 minutes of cool down.
  Interventions: Other: Thai dance with twenty-five squares (TDT)
- Control (CON) (Sham Comparator): The CON group did not have any intervention but usual care.
  Interventions: Other: Control (CON)

INTERVENTIONS:
Other: Thai dance with twenty-five squares (TDT) — The participants received a Thai dance with twenty-five squares (TDT) program 3 days/week, 12 weeks. This training comprises 10 minutes of warm up, following by 40 minutes of exercise at 40-50% of heart rate reserve at week 1-4, 50-60% of heart rate reserve at week 5-8, and 60-70% of heart rate reserve at week 9-12, 5 minutes of cool down.
  Arms: Thai dance with twenty-five squares (TDT)
Other: Control (CON) — The CON group did not have any intervention but usual care.
  Arms: Control (CON)

SUMMARY:
The objective of this study was to determine the effects of Thai dance with twenty-five squares on cerebrovascular and cognitive function in elderly with mild cognitive impairment

DETAILED DESCRIPTION:
Twenty elderly with mild cognitive impairment aged 60 years and over were randomized into 2 groups: control group (CON; n=20) and Thai dance with twenty-five squares training group (TDT; n=20). Participants in CON group do their daily routine without receiving any training program, while those in TDT group completed receiving Thai dance with twenty-five squares training program three time a week for twelve week-long (60 minutes/time). The physiological data, cerebrovascular function, cognitive, respiratory function, health-related physical fitness, and Blood biochemistry variables were analyzed during the pre-test and post-tests. The dependent variables between pre-test and post-tests were analyzed by paired t-test. The variables between pre-test and post-test were analyzed by paired t-test. In addition, an independent t-test was used to compare the variables between groups. Statistical significance was defined as p < .05.

ELIGIBILITY:
Inclusion Criteria:

* Elderly males and females aged 60-79 years who can lead normal daily lives. Individuals with mild cognitive impairment identified through the Montreal Cognitive Assessment (MoCA) with a score in the range of 17 - 25.
* Must be able to listen, speak, read, write, and understand the Thai language.
* Should not have diseases or abnormalities such as heart disease, eye complications caused by diabetes, uncontrolled high blood pressure, kidney complications caused by diabetes, and stroke.
* Must not have other respiratory diseases such as tuberculosis (Tuberculosis), asthma (Asthma), lung cancer (Lung cancer), emphysema (Emphysema), chronic obstructive pulmonary disease (COPD), etc.
* Must be a person not at risk of falling, determined through a test of the ability to walk and turn 3 meters within a time period of 7 - 15 seconds.
* Must not have received medication to treat dementia.
* Should not have received exercise training for more than 20 minutes at a time, 3 days/week, or more in the past 6 months before participating in the research.
* Should not have symptoms of mental disorders such as schizophrenia, bipolar disorder, or depression.
* Should have passed the pre-exercise readiness assessment (PAR-Q).
* Must be willing to participate in the research and sign the consent form to take part in the study.

Exclusion Criteria:

* A force majeure event, such as illness, that prevents participation in the research.
* Participation in less than 80% of the research sessions (must participate 29 times out of 36 times).
* Unwillingness to continue participating in the research.

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Cerebrovascular reactivity | Change from baseline Cerebrovascular reactivity at 12 weeks.
  Cerebrovascular reactivity is a test that assesses the response of cerebral blood vessels to carbon dioxide. This test analyzes the ability of cerebral blood vessels to contract and expand. Using an ultrasound machine and a probe with a frequency of 5 to 1 MHz, the partial pressure of CO2 is altered, and Cerebral Blood Flow Velocity (CBFV) is measured in the left middle cerebral artery at an examination depth of 30-65 mm. The variables used for analysis include Time-Averaged Peak Velocity (TAPV), Peak Systolic Velocity; PSV, End Diastolic Velocity; EDV, and Cerebral Blood Vessel Resistance (Pulsatility Index; PI).
Intima-Media Thickness (IMT) test | Change from baseline Intima-Media Thickness (IMT) at 12 weeks.
  Intima-Media Thickness (IMT) is a test conducted on the carotid artery on the side of the neck. Using an ultrasound machine (Philips, EPIQ 5G, USA), the thickness of the carotid artery walls was measured 1-2 cm away from the carotid bulb. Participants had their necks tilted 45 degrees. The artery walls were measured and then analyzed for thickness using the QLAB program.
Brachial-ankle pulse wave velocity (baPWV) | Change from baseline Brachial-ankle pulse wave velocity (baPWV) at 12 weeks.
  Brachial-ankle pulse wave velocity (baPWV) is utilized to indicate the arterial stiffness. This noninvasive test measure the time difference in blood pumping (brachial-ankle time delay) between the brachial artery and the posterior tibial artery. The length between both measurement points is then measured, and the pulse pressure wave between the upper arm and ankle is calculated (Brachial-ankle pulse wave velocity: baPWV), with the participant lying on their back on a bed. Next, both wrists and the left upper chest are cleaned with alcohol. The researcher then attaches cuffs to both the participants' arms and ankles, and electrodes of the device for measuring electrocardiograms are attached to the wrists. Additionally, cardiac sound waves (PCG) are placed on the left side near the sternum (Sternal notch).
Brain oxygen saturation levels | Change from baseline Brain oxygen saturation levels at 12 weeks.
  Brain oxygen saturation levels are assessed in the frontal lobe area using an oxygen saturation level meter (Universal Oximetry System), measured in percentage units. The evaluation is performed with a brain oxygen saturation level assessment device, specifically the SenSmart® Model X-100 (SenSmart® Model X-100, USA).
The Monreal Cognitive Assessment (MoCA-T) | Change from baseline MoCA-T scores at 12 weeks.
  The Monreal Cognitive Assessment, known as MoCA-T, is a questionnaire comprising 11 topics with a maximum score of 30 points. It serves as a comprehensive tool for assessing various aspects of cognitive intelligence in various areas, including management, naming, concentration, language use, and abstract thinking.
The Mini-Mental State Examination Thai (MMSE-T) | Change from baseline MMSE-T scores at 12 weeks.
  The Mini-Mental State Examination Thai (MMSE-T) is a preliminary brain condition test that comprises 11 topics with a maximum score of 30 points. This basic brain state test is utilized to assess various aspects of cognition, including awareness of surrounding conditions, perception of time, spatial orientation, concentration and calculation, language use, and repetition.
The Trail Making Test B Thai modified (TMT-B) | Change from baseline TMT-B testing time at 12 weeks.
  The Trail Making Test B Thai modified (TMT-B) is a subtest in the Halstead-Reitan Neuropsychological test, adapted into Thai. The criteria for normalcy is set at no more than 89 seconds for individuals aged 60 years and over. The test includes numbers 1-13 and month abbreviations in Thai (Jan. - Dec.), totaling 25 characters, which consist of numbers and/or letters. They are arranged in a distributed manner, and when connecting lines are drawn, they will not intersect. The TMT-B serves as an assessment of cognitive ability, focusing on concentration and management.

SECONDARY OUTCOMES:
Pulmonary function (Forced vital capacity; FVC) | Change from baseline FVC at 12 weeks.
  The participants were instructed to sit on a chair and wear a nose clip. The researcher provided them with a detailed set of instructions to ensure they performed the maneuver correctly according to guidelines of the American Thoracic Society (ATS). Prior to demonstrating forced inspiration and expiration, the participants were asked to perform three cycles of slow normal breathing as part of the FVC maneuver. FVC will be reported in liter (L).
Pulmonary function (Forced Expiratory Volume in one second; FEV1) | Change from baseline FEV1 at 12 weeks.
  The participants were instructed to sit on a chair and wear a nose clip. The researcher provided them with a detailed set of instructions to ensure they performed the maneuver correctly according to guidelines of the American Thoracic Society (ATS). Prior to demonstrating forced inspiration and expiration, the participants were asked to perform three cycles of slow normal breathing as part of the FVC maneuver. FEV1 (L) will be reported in liter (L).
Pulmonary function (The ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs; FEV1/FVC) | Change from baseline FEV1/FVC at 12 weeks.
  The participants were instructed to sit on a chair and wear a nose clip. The researcher provided them with a detailed set of instructions to ensure they performed the maneuver correctly according to guidelines of the American Thoracic Society (ATS). Prior to demonstrating forced inspiration and expiration, the participants were asked to perform three cycles of slow normal breathing as part of the FVC maneuver. FEV1/FVC will be reported in percent (%).
Pulmonary function (Maximal voluntary ventilation; MVV) | Change from baseline MVV at 12 weeks.
  The participants were instructed to sit on a chair and wear a nose clip. The researcher provided them with a detailed set of instructions to ensure they performed the maneuver correctly according to guidelines of the American Thoracic Society (ATS). During the MVV maneuver, participants were instructed to demonstrate in rapid and forceful inhalation and exhalation for a duration of 10 seconds. MVV will be reported in liter per minute (L/min).
Respiratory muscle strength | Change from baseline respiratory muscle strength at 12 weeks.
  Respiratory muscle strength was evaluated by measuring Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) in centimeters of water (cmH2O). The participants were seated and utilized a portable handheld mouth pressure meter (MicroRPM), along with a nose clip. To assess MIP, participants were instructed to exhale until they emptied their lungs at the point of functional residual capacity (FRC). Participants held the device to their mouth and forcefully inhaled for 1-2 seconds. For the measurement of MEP, participants were directed to inhale until their lungs were completely filled with air, starting from the total lung capacity (TLC) point. Participants were asked to maintain the device on their mouth and forcefully exhaled for 1-2 seconds.
The Chair Sit and Reach Test | Change from baseline The Chair Sit and Reach Test scores at 12 weeks.
  The Chair Sit and Reach Test is used to assess the flexibility of the back and legs. Participants sit in chairs with their feet touching the floor and positioned on the edge of the chair. The non-dominant leg should have the sole of the foot touching the floor, while the dominant foot is extended. Next, fold at the hips and reach with the middle finger of the hand on the same side as the outstretched leg to touch the middle finger to the outstretched foot. The researcher then measures the distance between the fingers and toes. If they touch each other, it indicates a distance equal to zero. Then, participants switch sides.
The Back Scratch test | Change from baseline The Back Scratch test scores at 12 weeks.
  The Back Scratch test is conducted to assess shoulder flexibility. Participants perform stretches targeting their shoulders, shoulder blades, chest, and arms, then stand upright. They lift their right arm above the shoulder, bend the elbow down behind the back in a palm-down position, with palms and fingers resting flat on the back. Participants press down as far as possible. Simultaneously, they raise their left arm backward in an inward twisting motion, bending the elbow and folding it up so that the backs of their hands rest against the back of their body. They lift their hands as high as possible, trying to bring the right and left hands together as much as possible. After holding for about 3 seconds, participants return to the starting position with arms released at their sides. The test is repeated two more times on each side. The assessment measures the distance between the tip of the middle finger of the upper hand and the tip of the radial styloid process of the lower hand.
The Time Up and Go test | Change from baseline The Time Up and Go test time at 12 weeks.
  The Time Up and Go test is a mobility and balance assessment. Participants begin by sitting in chairs with the soles of both feet touching the floor. At the start of the test, participants stand up, walk towards a target 3 meters from the starting point, circumnavigate the target, and then return to their original seat. The researcher measures the time from the starting point until the participant returns to a seated position.
The Chair Stand test | Change from baseline The Chair Stand test scores at 12 weeks.
  The Chair Stand test involves the use of a chair without armrests. The chair should be tall enough for participants to sit with their feet touching the floor. Initially, participants are asked to sit in the chairs. When the test begins, they stand up with both hands holding the shoulder blades in a crossed position. A timer is then set for 30 seconds to count how many times participants can sit and stand within that duration.
The Arm Curl test | Change from baseline The Arm Curl test scores at 12 weeks.
  The Arm Curl test involves participants holding a steel ball on their dominant side, weighing 5 pounds for women and 8 pounds for men. Participants lift the steel ball with their arms fully bent and stretch their arms as far as possible, counting as one repetition. Participants perform as many repetitions as possible within a 30-second time frame.
The 2-Minute Step Test | Change from baseline The 2-Minute Step Test scores at 12 weeks.
  The 2-Minute Step Test is an assessment of activity ability and endurance of the lower limb muscles. The researchers determined that the knee lift height for each elderly person would be at the midpoint between the knee and the upper edge of the hip bone. When the researcher gave the "start" command to the participants to raise their legs in place as many times as possible within 2 minutes, the researchers counted the number of leg lifts when the knees reached the designated point.
The 6-Minute Walk Test | Change from baseline The 6-Minute Walk Test scores at 12 weeks.
  The 6-Minute Walk Test is a sub-maximal exercise test used to assess the ability to perform activities for extended periods. Participants are instructed by the researcher to walk at their comfortable speed for 6 minutes, covering a minimum distance of 15 meters before turning around. The researcher records the distance walked within the 6-minute timeframe.
Blood chemical data test | Change from baseline blood chemical data at 12 weeks.
  Draw 15 milliliters of blood to analyze blood biochemistry, including fasting plasma glucose (FPG), accumulated blood sugar level (HbA1c), insulin resistance (Homeostasis Model Assessment; HOMA-IR), cholesterol (Cholesterol), high-density lipoprotein (HDL), low-density lipoprotein (LDL), triglycerides (Triglyceride), BDNF (Brain-Derived Neurotrophic Factor), interleukin-6 (IL-6), interleukin-10 (IL-10), and tumor necrosis factor-alpha (TNF-α).

CONTACTS AND LOCATIONS:
Overall Officials: Wannaporn Tongtako, Ph.D., Principal Investigator — Chulalongkorn University
Locations (2):
- Thailand (2):
  - Faculty of Sports Science, Chulalongkorn University, Pathum Wan, Bangkok
  - Wannaporn Tongtako, Bangkok

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Akazawa N, Tanahashi K, Kosaki K, Ra SG, Matsubara T, Choi Y, Zempo-Miyaki A, Maeda S. Aerobic exercise training enhances cerebrovascular pulsatility response to acute aerobic exercise in older adults. Physiol Rep. 2018 Apr;6(8):e13681. doi: 10.14814/phy2.13681. PMID 29687959
- [Result] Bherer L. Cognitive plasticity in older adults: effects of cognitive training and physical exercise. Ann N Y Acad Sci. 2015 Mar;1337:1-6. doi: 10.1111/nyas.12682. PMID 25773610
- [Result] Boyle PA, Buchman AS, Wilson RS, Leurgans SE, Bennett DA. Physical frailty is associated with incident mild cognitive impairment in community-based older persons. J Am Geriatr Soc. 2010 Feb;58(2):248-55. doi: 10.1111/j.1532-5415.2009.02671.x. Epub 2010 Jan 8. PMID 20070417
- [Result] Miller SM, Taylor-Piliae RE. Effects of Tai Chi on cognitive function in community-dwelling older adults: a review. Geriatr Nurs. 2014 Jan-Feb;35(1):9-19. doi: 10.1016/j.gerinurse.2013.10.013. Epub 2013 Oct 24. PMID 24252560